CLINICAL TRIAL: NCT01071590
Title: The Influence of Sensory Stimuli on Gait Imagery in Patients With Freezing of Gait
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100057; 10-N-0057
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2014-01-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Sensory Input; Gait; Imagery; Parkinson Disease; PD
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Freezing of gait (FOG) is a common and very disabling symptom in people with Parkinson s disease, significantly affecting their quality of life. It has been defined as a sudden break or block in the walking motion, or as an inability to start walking. Although certain neural connections or neurological processes might contribute to FOG, more research is needed to produce consistent findings. Researchers are interested in investigating brain function involved in FOG.

Objectives:

- To obtain more information on brain function in individuals with freezing of gait.

Eligibility:

* Individuals between the ages of 45 and 80 who have been diagnosed with Parkinson s disease.
* Participants must be willing to go off their current Parkinson s disease medications for up to 12 hours at a time.

Design:

* Participants will be divided into two groups: those who do have freezing of gait (more than about once a day) and those who have not experienced this symptom.
* The study will involve a screening visit (1 hour) and a study visit (2 hours).
* During the screening visit, participants will be asked about medical history, and will have physical, neurological, memory, and walking tests.
* Participants should not take their Parkinson's disease medications for 12 hours before the study visit. Participants who cannot come to the clinic safely without their medications will be allowed to stay in the hospital overnight before the visit, and should bring their medications to the study in order to take them as soon as needed after the study.
* Participants will be asked to perform several tasks before the imaging study: (1) walking 10 yards back and forth down a hallway, (2) walking 10 yards back and forth while following horizontal lines on the floor, (3) walking 10 yards back and forth while listening to a metronome, and (4) being pushed back and forth in a wheelchair.
* After participants perform the actual tasks, participants will be asked to imagine performing the tasks and fill out questionnaires about how well they can imagine the tasks.
* Participants will be monitored with a functional magnetic resonance imaging (fMRI) scan while imagining the four tasks they have just performed.

DETAILED DESCRIPTION:
Objective

Freezing of gait (FOG) is a common and very disabling symptom in Parkinson s disease (PD). It has been defined as a sudden transient break (motor block) in the walking motion or as an inability to generate effective stepping. It significantly affects PD patients, resulting in a decline in Quality of Life (QOL). Although certain neural substrates or neuronal connectivity might contribute to FOG, no consistent findings have been established. Our major goal is to investigate the pathophysiology of the brain as it relates to FOG.

Study population

We intend to study 46 PD patients (23 with freezing and 23 without).

Design

Assuming that certain neural networks or brain regions are associated with FOG, we are planning to investigate its mechanism by measuring the Blood Oxygen Level Dependent (BOLD) effect with functional MRI (fMRI) during motor imagery (MI) of gait in PD patients with and without FOG, and compare the results with each other.

Using a block design in functional magnetic resonance imaging (fMRI), we will examine brain activity and brain connectivity of PD patients with and without freezing while they execute four tasks: normal gait imagery; gait imagery with lines on the floor (visual cue); gait imagery with sounds of the metronome (auditory cue); and imagery of being moved by the experimenter while sitting in a wheelchair. The last condition is done to control for the visual flow which should be experienced during MI of gait.

It is known that the motor ability of PD patients, both those with and without FOG, improves with exposure to certain visual stimuli. Using a treadmill combined with a virtual reality environment, we will test the effect of different visual stimuli on the gait performance of PD subjects with and without FOG. In particular, we will examine gait performance as it relates to FOG.

Outcome Measures

For the fMRI experiment, the primary outcome measure is the change of BOLD-MRI signals and the functional connectivity of the activated regions during different conditions and between groups. In addition, the Vividness of Movement Imagery Questionnaire (VMIQ) score (Isaac A, 1986) will also be collected as a secondary outcome measure.

Another secondary outcome measure involves the treadmill experiment. In this test, the outcome measure is the motion analysis data, such as stride length and speed, which are derived from the VICON system. Using this test, we hope to determine when the FOG phenomenon occurred.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. PD patients with freezing:

     1. 40 to 80 years of age with idiopathic PD
     2. Hoehn and Yahr stage 1-4
     3. Answer to the FOGQ item 3 range from 3-4 (freezing more than about once a day).
     4. Existence of FOG documented by a neurologist
     5. Currently taking medications for PD such as L-DOPA (Sinemet) or dopamine agonists such as Mirapex or ReQuip.
     6. Willing and able to be off your PD medications for at least 12 hours for visit 1 and visit 2.
  2. PD patients without freezing:

     1. 40 to 80 years of age with idiopathic PD
     2. Hoehn and Yahr stage 1-4
     3. Answer to the FOG item 3 is 0 (Never freezes).
     4. The lack of existence of FOG documented by a neurologist.
     5. Currently taking medications for PD such as L-DOPA (Sinemet) or dopamine agonists such as Mirapex or ReQuip.
     6. Willing and able to be off your PD medications for at least 12 hours on one occasion.

Patients in the FOG group and the non-FOG group will be matched by clinical disease stage.

EXCLUSION CRITERIA:

1. Any active psychiatric disease or evidence of dementia
2. Feel uncomfortable being in small, enclosed spaces (claustrophobia) or unable to lie still for an hour, e.g. due to back pain
3. Pallidotomy or implanted electrodes and generator for deep brain stimulation
4. Pregnancy
5. Surgically or traumatically implanted foreign bodies such as a pacemaker, implanted medical pump, implanted hearing aids, metal plate in the skull, or metal implant in the skull or eyes (other than dental appliances or fillings) that may pose a physical hazard during MRI.
6. Inability to provide informed consent
7. Unable to walk a 10 meter distance even with help of an assisting device
8. Unable or unwilling to withhold PD medications for 12 hours prior to visit 1 and visit 2
9. Have a neurologic condition other than PD, such as a brain tumor, stroke, head trauma or a vascular malformation
10. Have a dysfunction of vision, such as severe loss of visual acuity, that impairs his/her ability to perform the visual imagery task or to appreciate the virtual reality environment during the treadmill test

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-02-01; Study Completion 2014-01-03

PRIMARY OUTCOMES:
The change of BOLD-MRI signals and the functional connectivity of the activated regions during different conditions and between groups

SECONDARY OUTCOMES:
Vividness of Movement Imagery Questionnaire (VMIQ) score (Isaac A, 1986) will also be collected as a secondary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Atchison PR, Thompson PD, Frackowiak RS, Marsden CD. The syndrome of gait ignition failure: a report of six cases. Mov Disord. 1993 Jul;8(3):285-92. doi: 10.1002/mds.870080306. PMID 8341292
- [Background] Azulay JP, Mesure S, Amblard B, Blin O, Sangla I, Pouget J. Visual control of locomotion in Parkinson's disease. Brain. 1999 Jan;122 ( Pt 1):111-20. doi: 10.1093/brain/122.1.111. PMID 10050899
- [Background] Bartels AL, Leenders KL. Brain imaging in patients with freezing of gait. Mov Disord. 2008;23 Suppl 2:S461-7. doi: 10.1002/mds.21912. PMID 18668627